CLINICAL TRIAL: NCT05502757
Title: Fresh Fruits and Vegetables for Families (or Fresh Families) Study
Brief Title: Fruit & Vegetable Provision Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators decided not to move forward with study.
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Associate Dean of Research, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UTK IRB-22-06985-XP
Record Dates: First submitted 2022-08-02; First posted 2022-08-16 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Food Security
Keywords: Food provision
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provision of paper FV vouchers (VOUCHER) condition (Experimental): Families in the VOUCHER condition will be provided 6, $15 paper vouchers ($90 total) for the purchase of fresh FV at a partnering Food City location in Knoxville, TN.
  Interventions: Other: Fruit and vegetable provision
- Home delivery of fresh FV (DELIVERY) condition (Experimental): Families in the DELIVERY condition will be provided access to an online Food City account to purchase up to $90 fresh FV for home delivery, delivered by research staff at the time of their choosing.
  Interventions: Other: Fruit and vegetable provision

INTERVENTIONS:
Other: Fruit and vegetable provision — Fresh fruits and vegetables are provided to families at no cost

SUMMARY:
Fresh Families is a research study being conducted by the Healthy Eating and Activity Laboratory at the UT Dept of Nutrition. The purpose of this study is to see which food provision strategy, paper vouchers or home delivery, best increases fruit and vegetable (FV) availability at home and child FV intake. The study will enroll families experiencing household food insecurity with children 4-17 years who do not meet recommendations for FV intake and have an adult caregiver (18+ years) willing to participate. Families will be randomized to one of two groups: voucher group or home delivery group. Families in the voucher group will be provided 6, $15 paper vouchers ($90 total) for the purchase of fresh FV at a partnering Food City location in Knoxville, TN. Families in the home delivery group will be provided access to an online Food City account to purchase up to $90 fresh FV for home delivery, delivered by research staff at the time of their choosing. Each group will have 6 weeks to utilize their vouchers/funds, and then they will expire. There will also be one appointment to collect child and caregiver height and weight at the family's home.

DETAILED DESCRIPTION:
Purpose/objectives of the study

Research has shown that children experiencing food insecurity are not meeting recommended intake of fruits and vegetables (FV). Cost and transportation/geographical barriers to accessing FV may be barriers that prevent these children from consuming recommended amounts of FVs. Food provision strategies, such as FV delivery or vouchers, may mitigate these barriers, assisting with increasing FV intake. Thus, efficacious strategies for food provision are needed for families with children who are experiencing food insecurity.

The purpose of this study is to see which food provision strategy, paper vouchers or home delivery, best increases FV availability at home and child FV intake.

Recruitment

For recruitment, flyers will be provided to interested elementary schools, daycare centers, Head Start locations, and community organizations within the 5-mile radius of the Western Ave Food City store. According to each organization's preference, paper flyers to hang and/or digital flyers to be distributed via listservs and/or social media will be provided. Flyers and listservs will also be used on the UTK and UTIA campuses, and study advertisements will be launched on Facebook. Additionally, summer meal sites (https://www.fns.usda.gov/meals4kids) will be contacted within the 5-mile radius to ask permission to handout study flyers at these events. Additionally, research staff will also set up recruitment tables at relevant family and community events, children's events and festivals, and health fairs in this zone. Recruitment flyers/advertisements will display a QR code that interested parents can scan using the camera app on their smartphone. The QR code will direct the parent to a brief Qualtrics survey that asks a few screening questions, collects contact information (caregiver name, phone number, and email), and obtains permission to be contacted by the research staff. Interested families will be contacted by the research team and screened for eligibility by phone. Eligible families will be then invited to an orientation. These orientations will be conducted virtually over Zoom. The orientations sessions will occur one-on-one between a family and a research team member. Families will be mailed/emailed the consent forms prior to the orientation. For families who are interested, the research team will review the consent form at the end of the orientation, and adult caregivers will sign consent forms and children will provide assent (verbal or written). Consent/assent forms will be collected via Qualtrics.

Study/Project Procedures

This study will utilize a randomized experimental design. After completion of consent/assent procedures, families will complete a baseline assessment (see Baseline Assessment section below), and then be randomized to one of two 6-week programs using a random numbers table: 1) provision of paper FV vouchers (VOUCHER) or 2) home delivery of fresh FV (DELIVERY). Research staff will then provide instructions for purchasing FV based on randomization condition. For the instructions, families in the VOUCHER condition will be informed of the process for making FV purchases with paper vouchers in the partnering grocery store. For families in the DELIVERY condition, research staff will share their screen on Zoom to demonstrate how to navigate the online food ordering process on the Food City website. Families will be provided with electronic documents regarding instructions for their condition at this session.

Within 2 days of the assessment, a home visit will occur in which families in both conditions will be provided with hard-copy materials covering instructions for their randomized condition, as well as basic nutrition education materials on FV and a community resource guide. At this time, the VOUCHER condition will receive their paper vouchers and the DELIVERY condition will be provided access to an online Food City account maintained by the research staff along with delivery windows for the upcoming week. To reduce participant burden, research staff will attempt to schedule the height and weight measure (se Baseline Assessment section below) at this same home visit. If that can't occur, an additional home visit will be scheduled for these measure, with this visit occurring within two weeks of the assessment.

Families will have a period of 6 weeks to redeem their FV benefits, and follow-up measures will be collected during week 5 of the purchasing period. Including the orientation/baseline Zoom visit, study length will be just over 8 weeks in duration.

Provision of paper FV vouchers (VOUCHER condition)

For families in the VOUCHER condition, paper vouchers will be hand-delivered within 2 days after baseline assessment. Date of delivery will mark the beginning of the 6-week purchasing period for the FV vouchers. Participants can use these vouchers to purchase fresh FV at our retail grocery partner Food City, located at 1950 Western Ave., Knoxville, TN, 37921. The families will receive 6, $15 vouchers ($90 total), or approximately $1 per day for the participating child and caregiver. Vouchers may only be used once, meaning that if there is any unused value left on the voucher, it will be lost. Families can use the vouchers in whatever manner is appropriate for them over the six weeks (e.g., all at once, one every week, etc). The vouchers will expire 6 weeks from the date they are delivered. Families will receive text messages at the end of weeks 1-5 to remind them to use the vouchers. At the end of week 5, the text will also include a reminder that the vouchers expire in one week. If a family reports one or more vouchers as lost, they will be issued new vouchers.

Home delivery of fresh FV (DELIVERY condition)

As in the VOUCHER condition, participants in the DELIVERY condition will be allotted up to $90 in fresh FV purchases. Participants will be provided access to an online Food City account maintained by the research staff beginning 2 days after baseline assessment. Access to online delivery will expire 6 weeks from this date. Prior to deliveries, families will fill a virtual cart with their preferred fresh FV. To mimic the VOUCHER condition, purchases in the DELIVERY condition will also be subject to the $15-increment rule (i.e., unused funds up to the next $15-increment will be considered lost). Similar to the vouchers, families can use the $90 in whatever manner is appropriate for them over the six weeks (e.g., all at once, $15 increments every week, etc). To ensure that only fresh FV are purchased, and in the correct amount, families will be required to fill their carts at least one day before their desired delivery time. This will provide time for research staff to review the purchases and provide feedback, if needed. Families will send a text to the lab phone by close of business (5:00 PM) on the day prior to delivery to indicate their order is complete and ready for review, and research staff will respond with a confirmation text. If there is an issue with the cart (exceeds voucher limit, includes items other than FV, etc.), research staff will follow-up with the family until the order is finalized.

Food City employees will shop for online orders according to their regular business model and/or UTK student research assistants will shop for the ordered items at the partner Food City location. Sometimes items listed as available online may be out-of-stock in the store. To ensure participants are able to redeem the full value they intended, families will provide a preferred list of fresh FV that can be substituted for out-of-stock items. These preferred items will be included in a note to the Food City shopper in the online system that indicates he/she should replace out-of-stock items with an equivalent value of a participant's preferred FV.

Families will be able to choose a convenient delivery time from pre-specified delivery windows determined by research staff availability. Each week, families will receive a text reminder that lists the available windows for grocery delivery. Since families in the VOUCHER condition will not have a tangible reminder of remaining money for FV purchases (i.e., physical paper vouchers), study staff will track purchases over time. Text messages will include reminders of the family's remaining balance. When the $90 limit is reached, text message reminders will cease. The morning of the delivery, participants will receive a text message reminder. A research staff member will deliver the groceries to the participant's home during the scheduled window, following any health safety procedures in place at the time, and will make a good faith effort to hand the groceries off to the family. However, if the family cannot be contacted or is not home during the time of the scheduled delivery, the groceries will be left on the participant's doorstep in cold storage bags.

Baseline Assessment

Baseline assessment will occur via Zoom. Following the signing of the Qualtrics consent/assent forms, research staff will provide families a link to complete baseline assessment questionnaires via Qualtrics. Parent and child height and weight measures will occur within 2 weeks of baseline assessment and collected in person by research staff, following health safety procedures that may be in place.

Post-Intervention Assessment

Follow-up assessments will occur during week 5 of the purchasing period. Families will be sent a link to the follow-up assessment questionnaires on Qualtrics. A unique survey link will be created for each family so that responses can be matched to the participant.

ELIGIBILITY:
Inclusion Criteria:

* Families experiencing food insecurity
* Live within a 5-mile radius of the partnering Food City location
* Have a child 4 to 17 years of age
* Adult (> 18 years) caregiver living in the household willing to participate in the program will be eligible
* Adult caregiver must be able to read and speak English
* Adult caregiver willing to shop for fresh FV at the partnering Food City location

Exclusion Criteria:

* Families with children who currently meet current recommendations for FV intake (i.e., ≥4.5 cups of FV/day, based on Dietary Guideline for Americans 2020-2025 Healthy US-Style Dietary Pattern for Ages 2 and Older)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Total spent on fruits and vegetables (both groups) | 6 weeks
  For the VOUCHER group, research staff will work with the partner Food City to determine total amount spent on fresh fruits and vegetables using vouchers. For the DELIVERY group, research staff will retain all grocery receipts to determine the total amount used. (Up to $90 for both groups.)
Number of vouchers used (VOUCHER group only) | 6 weeks
  Total number of vouchers used by the participant
Average amount of voucher value used (VOUCHER group only) | 6 weeks
  The average amount of money used from each voucher (up to $15 per voucher)
Purchase amount per delivery (DELIVERY group only) | 6 weeks
  The average purchase amount spent for each delivery

SECONDARY OUTCOMES:
Child BMI z-scores | Baseline only
  Child height and weight will be used to calculate child BMI z-scores using the CDC BMI-for-age charts, 2 to 20 years, by sex and age
Caregiver BMI | Baseline only
  Caregiver weight and height will be combined to report BMI in kg/m^2
Demographics | Baseline only
  Demographics will be assessed and used to describe the study sample. Demographics collected will include child and caregiver measures of age, gender, race/ethnicity, and caregiver measures of marital status, caregiver education level, employment status, and income.
Household information | 6 weeks
  The number of people living in the household and federal food program participation (like SNAP, WIC, school breakfast and lunch) will be collected.
Fruit and vegetable purchases | 6 weeks
  The Food Purchasing and Household Food Availability survey will be used to determine whether common fruits and vegetable items have been purchased for the household in the last month.
Fruit and vegetable home availability | 6 weeks
  The Food Purchasing and Household Food Availability survey will be used to determine if common fruits or vegetable items are available at the time of survey administration.
Food Security | 6 weeks
  Food security will be assessed using the gold-standard USDA food security modules to test for food insecurity in both adults and children in a household. Scores will be compared pre to post intervention to determine if provision of the fruit and vegetable prescription vouchers/home deliveries aided families in accessing more food/reducing their level of food insecurity.
Fruit and Vegetable Dietary Screener | 6 weeks
  he National Cancer Institute's fruit and vegetable dietary screener will be administered to child participants to determine if there are changes in dietary intake of fruits and vegetables before and after the provision of vouchers/home deliveries. This screener will be completed for the child participant by the adult caregiver.
Food Attitudes and Behaviors | At 6-week follow-up only
  The National Cancer Institute's FAB questionnaire will be administered to parents to determine whether they experience some common barriers to eating fruits and vegetables.
Satisfaction Survey | At 6-week follow-up only
  A short survey will be administered at the post-intervention assessment to obtain participant feedback on their satisfaction with and perceptions of their assigned food provision method (VOUCHER vs DELIVERY).
Types of fruits and vegetables purchased | 6 weeks
  Using receipt and voucher data, research staff will examine the types of fresh fruits and vegetables purchased by participants in each group (VOUCHER vs DELIVERY)

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD RD LDN, Principal Investigator — University of Tennessee Knoxville, Department of Nutrition
Locations (1):
- Healthy Eating and Activity Lab, University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haynes-Maslow L, Parsons SE, Wheeler SB, Leone LA. A qualitative study of perceived barriers to fruit and vegetable consumption among low-income populations, North Carolina, 2011. Prev Chronic Dis. 2013;10:E34. doi: 10.5888/pcd10.120206. PMID 23489639
- [Background] Bihan H, Mejean C, Castetbon K, Faure H, Ducros V, Sedeaud A, Galan P, Le Clesiau H, Peneau S, Hercberg S. Impact of fruit and vegetable vouchers and dietary advice on fruit and vegetable intake in a low-income population. Eur J Clin Nutr. 2012 Mar;66(3):369-75. doi: 10.1038/ejcn.2011.173. Epub 2011 Oct 12. PMID 21989324
- [Background] Jones LJ, VanWassenhove-Paetzold J, Thomas K, Bancroft C, Ziatyk EQ, Kim LS, Shirley A, Warren AC, Hamilton L, George CV, Begay MG, Wilmot T, Tsosie M, Ellis E, Selig SM, Gall G, Shin SS. Impact of a Fruit and Vegetable Prescription Program on Health Outcomes and Behaviors in Young Navajo Children. Curr Dev Nutr. 2020 Jul 21;4(8):nzaa109. doi: 10.1093/cdn/nzaa109. eCollection 2020 Aug. PMID 32734135
- [Background] Locher I, Waselewski M, Sonneville K, Resnicow K, Chang T. Grocery Delivery of Healthy Foods to Pregnant Young Women With Low Incomes: Feasibility and Acceptability Mixed Methods Study. JMIR Form Res. 2020 Dec 24;4(12):e21602. doi: 10.2196/21602. PMID 33361055

DOCUMENTS (1):
  • Informed Consent Form (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT05502757/ICF_001.pdf